CLINICAL TRIAL: NCT06961500
Title: A Multicenter, Phase 2, Randomized Trial of Obinutuzumab With CHOP Versus Obinutuzumab With Bendamustine in the Treatment of Newly Diagnosed Follicular Lymphoma Grade 3A (FL)
Brief Title: Obinutuzumab With CHOP Versus Obinutuzumab With Bendamustine in the Treatment of Newly Diagnosed Follicular Lymphoma Grade 3A
Acronym: PROOF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-125-01
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Follicular Lymphoma Grade 3A
MeSH Terms: interventions — obinutuzumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obinutuzumab and CHOP Combination Treatment (Active Comparator): Obinutuzumab: 1000mg i.v., administered on Day 1/8/15 (D1/8/15) of Cycle 1 (C1), and D1 of C2-6.
  CHOP: a) Cyclophosphamide: 750 mg/m2 i.v. drip, administered on D1; b) Doxorubicin: 50 mg/m2 i.v. drip (or Epirubicin: 70mg/m2 i.v. drip), administered on D1; c) Vincristine: 1.4 mg/m2 i.v., administered on D1; d) Prednisone: 100mg/d po, administered on D1-5.
  Each cycle lasts 21 days, up to 6 cycles are administered. Then add 2 cycles of obinutuzumab monotherapy.
  Interventions: Drug: Obinutuzumab; Drug: CHOP
- Obinutuzumab and Bendamustine Combination Treatment (Experimental): Obinutuzumab: 1000mg i.v., administered on D1/8/15 of C1, and D1 of C2-6. Bendamustine: 90 mg/m2 i.v. drip, administered on D1-2. Each cycle lasts 28 days, up to 6 cycles are administered.
  Interventions: Drug: Obinutuzumab; Drug: Bendamustine

INTERVENTIONS:
Drug: Obinutuzumab — 1000mg i.v., administered on Day 1/8/15 (D1/8/15) of Cycle 1 (C1), and D1 of C2-6
Drug: CHOP — a) Cyclophosphamide: 750 mg/m2 i.v. drip, administered on D1; b) Doxorubicin: 50 mg/m2 i.v. drip (or Epirubicin: 70mg/m2 i.v. drip), administered on D1; c) Vincristine: 1.4 mg/m2 i.v., administered on D1; d) Prednisone: 100mg/d po, administered on D1-5.
  Arms: Obinutuzumab and CHOP Combination Treatment
Drug: Bendamustine — 90 mg/m2 i.v. drip, administered on D1-2.
  Arms: Obinutuzumab and Bendamustine Combination Treatment

SUMMARY:
This is a multicenter, phase 2, randomized trial to evaluate the efficacy and safety of obinutuzumab with CHOP versus obinutuzumab with bendamustine in treatment-naïve follicular lymphoma (Grade 3A) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed follicular lymphoma Grades 3A, CD20 positive by immunohistochemistry.
2. Meets at least one GELF (Groupe d'Etude des Lymphomes Folliculaires) criteria.
3. No prior systemic treatment for lymphoma.
4. Presence of measurable lesions.
5. Age ≥ 18 years, no gender restriction.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. Expected survival of > 3 months.
8. Adequate organ and bone marrow function.

Exclusion Criteria:

1. History of allergy to any component of monoclonal antibodies or investigational drugs.
2. Central nervous system involvement.
3. History of previous malignant tumors.
4. History of active bleeding or bleeding tendencies, or requiring anticoagulant medication.
5. Requirement for potent CYP3A4 inhibitors for treatment.
6. Active infection, except for tumor-related B symptoms.
7. Known history of Human Immunodeficiency Virus (HIV) infection and/or acquired immunodeficiency syndrome (AIDS).
8. Hepatitis C virus (HCV) antibody positive with HCV RNA quantitative test result exceeding the detection limit; Hepatitis B surface antigen (HBsAg) positive or Hepatitis B core antibody (HBcAb) positive, with Hepatitis B virus DNA quantitative test result exceeding the detection limit (for patients with HBsAg or HBcAb positive status, regardless of HBV-DNA detection, oral entecavir or other antiviral therapy must be initiated prior to enrollment and continued according to the physician's instructions during the trial).
9. Significant organ dysfunction or uncontrolled comorbidities, such as uncontrolled hypertension, decompensated cirrhosis, uncontrolled diabetes, chronic obstructive pulmonary disease, etc.
10. History of severe heart disease.
11. Major surgery within 4 weeks prior to enrollment.
12. Participation in other clinical trials with drug intervention within 4 weeks prior to enrollment.
13. Pregnant or breastfeeding women, or planning to become pregnant during the study.
14. Individuals with psychiatric disorders, history of alcohol or drug abuse, or inability to provide informed consent.
15. Investigator determines the patient is unsuitable for enrollment or may not be able to complete the trial for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Assessed up to 5 years.
  From study entry to the first documented disease progression or death from any cause.

SECONDARY OUTCOMES:
Complete Response (CR) | Up to 6 cycles (up to 24 weeks).
  Defined as the proportion of patients who achieve complete remission at the end of induction therapy.
Objective Response Rate (ORR) | Up to 6 cycles (up to 24 weeks).
  The proportion of patients who achieve complete remission (CR) or partial remission (PR) at the end of induction therapy.
Event-Free Survival (EFS) | Assessed up to 5 years.
  From study entry to the first occurrence of any event, including disease progression, discontinuation of treatment, or death for any reason.
Overall Survival (OS) | Assessed up to 5 years.
  From study entry to death from any cause.
Progression of Disease within 24 months (POD24) | 24 months.
  The occurrence of disease progression or relapse within 24 months from the date of enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided